CLINICAL TRIAL: NCT07397507
Title: Mechanisms of Written Exposure Therapy in Residential SUD Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Robyn Ellis, Clinician Investigator, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P003371
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: PTSD - Post Traumatic Stress Disorder; Substance Use Disorder (SUD)
Keywords: PTSD treatment; Written Exposure Therapy; Substance Use Disorder; treatment mechanisms; fear extinction
MeSH Terms: conditions — Combat Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WET (Experimental): This arm will receive Written Exposure Therapy in addition to residential SUD treatment.
  Interventions: Behavioral: Written Exposure Therapy
- Neutral Writing (Other): This arm will receive five sessions of neutral writing in addition to residential SUD treatment.
  Interventions: Behavioral: Neutral Writing

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Written Exposure Therapy (WET) is a five-session manualized treatment for PTSD. At the first session, psychoeducation about common reactions to trauma and PTSD are presented followed by a 30-minute written exposure. Following the exposure, a 10-minute check-in is completed, and individuals are instructed not to avoid any thoughts/feelings/ images related to the trauma between sessions. All subsequent sessions follow this structure: check-in on avoidance and feedback on writing, written exposure, and brief check-in post-writing about the writing process.
  Arms: WET
Behavioral: Neutral Writing — Participants will complete five writing prompts that are not intended to provoke emotional responses. Examples of these prompts include writing about the food they ate the day prior or what they did yesterday. Participants will be instructed to not discuss their thoughts and feelings regarding these topics. Neutral writing will provide control for time and clinician contact.
  Arms: Neutral Writing

SUMMARY:
The goal of this clinical trial is to learn how Written Exposure Therapy (WET), a brief treatment for PTSD, works among individuals with substance use disorders (SUD) engaged in residential SUD treatment and how biology may influence treatment. The main questions it aims to answer are:

* Does WET improve PTSD and substance use outcomes among individuals with SUD+PTSD?
* Does WET improve physiological responses and craving to trauma cues?
* Do sex hormones influence changes physiological responses and craving during treatment among women?

Participants will:

* Complete WET or a neutral writing in addition to their residential SUD treatment
* Complete two laboratory sessions before and after treatment
* Complete follow-up surveys and interviews at 1- and 3-months post-treatment

ELIGIBILITY:
Inclusion Criteria:

1. ability to understand and sign informed consent
2. ability to write in English;
3. age between 18-55 (average age of menopause in the US)
4. [women only] naturally cycling (i.e., regular cycles, not on gonadal-related hormones)
5. current diagnosis of a moderate or severe DSM-5 SUD
6. current diagnosis of DSM-5 PTSD
7. sufficient memory of the trauma to write about the event
8. at least 5 business days left in their residential treatment episode (to allow for 5 treatment sessions).

Exclusion Criteria:

1. presence of a psychiatric or medical condition that would interfere with participation (e.g., severe, uncontrolled psychosis)
2. prescription of a PRN benzodiazepine
3. current PTSD treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptom Severity | Baseline, Immediately after intervention, 1- and 3-Month Post-Discharge
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure of symptoms of PTSD as defined by the DSM-5. Participants are instructed to keep in mind the identified worst event when responding to the items. Items are summed to create a total score which ranges from 0-80; a total score cut-off of 33 is recommended for identifying probable PTSD.
Days of Substance Use | Baseline, 1- and 3-Month Post-Discharge
  The Timeline Follow-Back (TLFB) method will be used to assess past 30-day substance use frequency and quantity. The TLFB will be administered by phone at 1-month and 3-month post-discharge. Days of use at Baseline will ask about the 30 days prior to entering treatment.
Heart Rate (HR) | Baseline, Intervention Sessions, Immediately after intervention
  Biopac MP150 for Windows will be used to collect electrocardiogram (ECG) data at a sampling rate of 1000 Hz. ECG is measured using three disposable Ag/AgCl electrodes and data are processed using MindWare software. HR will be derived by spectral analysis of 1-min epochs with a Hamming windowing function and log transformed. HR will be measured continuously during the trauma-cue reactivity paradigm (primary outcome), and during WET treatment sessions (secondary outcome). Average HR in beats per minute will be calculated during the trauma-cue (primary) and for each 30-minute writing session (secondary).
Skin Conductance Response (SCR) | Baseline, Intervention Sessions, Immediately after intervention
  Biopac MP150 for Windows will be used to collect electrodermal activity (EDA) data at a sampling rate of 1000 Hz. EDA is measured using two finger electrodes and data are processed using MindWare software. EDA will be measured continuously during the trauma-cue reactivity paradigm (primary outcome), and during WET treatment sessions (secondary outcome). SCR will be calculated as the maximum SC amplitude during the trauma-cue adjusted for the average SC amplitude during the final 30-seconds of the rest phase (primary outcome). SCR during each WET session (secondary outcome) will be calculated as the maximum EDA amplitude during the written exposure, adjusted for baseline amplitude.
High-Frequency Heart Rate Variability (HF-HRV) | Baseline, Intervention Sessions, Immediately after intervention
  Biopac MP150 for Windows will be used to collect electrocardiogram (ECG) data at a sampling rate of 1000 Hz. ECG is measured using three disposable Ag/AgCl electrodes and data are processed using MindWare software. HF-HRV will be derived by spectral analysis of 1-min epochs with a Hamming windowing function and log transformed. HF-HRV will be derived from ECG R-R intervals (inter-beat interval). Standard recommendations for the high frequency band settings (0.12- 0.40 Hz) will be used. HF-HRV will be measured during the trauma-cue reactivity paradigm (primary outcome), and during WET treatment sessions (secondary outcome). Average HF-HRV will be calculated during the trauma-cue (primary) and for each 30-minute writing session (secondary).
Trauma-Reactive Craving | Baseline, Intervention Sessions, Immediately after intervention, 1- and 3-Month Post-Discharge Follow-ups
  The Craving Scale is a 3-item validated measure of substance use craving. It uses a scale of 0-9 to assess: (1) the strength of craving in the past 24 hours, (2) the likelihood of use in an environment they have used in before, and (3) strength of cued craving. Craving will be assessed at all time points. Craving before and after the trauma-cue reactivity paradigm will be assessed and trauma-reactive craving will be the change in craving pre/post-trauma-cue (primary outcome). During the WET Intervention Sessions, substance use craving pre- and post- writing will be assessed and trauma-reactive craving will be calculated as post-writing craving adjusted for pre-writing craving (secondary outcome).

SECONDARY OUTCOMES:
Consequences of Substance Use | Baseline, Immediately after intervention, 1- and 3-Month Post-Discharge
  The Short Inventory of Problems - Revised (SIP-R) is a 17-item self-report of adverse consequences associated with drug or alcohol use in four domains: physical, social, intrapersonal, interpersonal, and impulse control. Items are rated on a scale of 0 (Never) to 3 (Daily or Almost Daily) representing the frequency of each consequence. A total score is calculated by summing all items, with higher scores reflecting greater consequences.